CLINICAL TRIAL: NCT05826314
Title: Impact of Boxing-based Training Program on Physical-functional Fitness, Cognitive Performance, and Risk of Falls in Community-dwelling Older Adults
Brief Title: Boxing Training, Physical-functional Fitness and Cognitive Performance in Older Adults
Acronym: Boxe4Ageing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Faculdade de Desporto da Universidade do Porto (Unknown); Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Lucimere Bohn, PhD, Universidade do Porto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262022
Record Dates: First submitted 2023-03-20; First posted 2023-04-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy People Programs
Keywords: Public health; Boxing; Elderly; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study includes a quasi-experimental design (non-randomized controlled trial), with repeated measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (adapted boxing) (Experimental): Experimental boxing - The general structure of adapted boxing will include a 10-minute warm-up consisting of walking at a slow, self-selected speed, and at the same time joint rotation exercises; followed by 25-30 minutes of adapted boxing (consisting of non-contact activities, distributed in coordination and balance/footwork, shadow boxing-choreography (sequence of arm and leg movements that simulate an imaginary fight and punching bag), to end the session there will be a content fixation exercise, relaxation with gentle movements and breathing for 5 -10 minutes.
  Interventions: Other: Boxing training
- Experimental group 2 (multi-component training) (Active Comparator): Sessions will be divided in 10 minutes warm-up (including slow walk, postural and mobility exercises for general activation, and stretching exercises), specific training (25-30 minutes, including balance/coordination training, strength, and aerobic exercises) and cool down 5 - 10 minutes (breathing and stretching exercises for the main worked joints and muscles) following the main guidelines recommended by the American College of Sports Medicine (4) and the WHO (3).
  Interventions: Other: Exercise
- Control group (No Intervention): Participants from the control group will participate in all assessments moments, and will be asked to maintain their usual activities. At the end of the intervention period, the control group will be invited to participate in a physical activity program that takes place at the University.

INTERVENTIONS:
Other: Boxing training — Training protocol will be held for 24 weeks, twice per week/ 45 min per sessions.
  Other Names: Combat sports
  Arms: Experimental group 1 (adapted boxing)
Other: Exercise — Training protocol will be held for 24 weeks, twice per week/ 45 min per sessions.
  Other Names: Multicomponent training
  Arms: Experimental group 2 (multi-component training)

SUMMARY:
The aim of the study is to evaluate and to compare the effects of two exercise regimes (Boxing Training -BT and Multicomponent Training -MT) and 12 weeks of follow-up on cognitive health status, physical-functional fitness, and risk of falls in community-dwelling elders.

This is a quasi-experimental controlled trial using a parallel-group design. Participants will be allocated to 3 groups (i.e. BT, MT or control group [no intervention]). Both exercise programs (BT and MT) will last 24 weeks, twice a week, 45 minutes per session. Participants of all groups will be assessed for Senior Fitness test, and body weight at 4 moments (baseline, 12 weeks and 24 weeks of exercise and a follow-up period lasting 12 weeks).

Our hypotheses are:

1. In comparison with the control group, both exercise groups (BT and MT) will positively improve their physical-functional fitness, cognitive health status and risk of falls with the interventions
2. The observed effects on physical-functional fitness, cognitive health status, and risk of falls as a result of the exercise programs will be similar.
3. During the follow-up period, both exercise groups will experiment reductions on physical-functional fitness, cognitive health status, and risk of falls.

DETAILED DESCRIPTION:
Aging is associated with functional and cognitive decline (1, 2), which are causal factors of falls in the elderly. According to available evidence, alleviation of these conditions can be achieved through regular exercise of the multicomponent type (MT) (3). However, in TM programs, "muscle power" takes a secondary role (5) although it is extremely important to preserve the integrity of the neuromuscular system (6). Studies indicate that combat sports may represent an exercise strategy that combines muscular fitness, cardiorespiratory fitness, agility, and balance (7), in addition to falling within the scope of dual-task programs (i.e., physical and cognitive) because they require memorization of combinations of attacking and defending movements, quick decision-making, and movement by coordinating simultaneous leg and hand movements (8). Seminal work with adapted boxing for elderly parkinsonians has demonstrated positive results in health indicators (9, 10). But the effectiveness of this modality in apparently healthy elderly is still unknown. Therefore, this project aims to compare the effects of boxing training and multi-component training on physical-functional fitness, cognitive performance, and the risk of falls in older people.

The study comprises a quantitative quasi-experimental design, will be conducted in the metropolitan area of Porto, Portugal. The study sample will consist of healthy individuals from the community, aged ≥ 60 years, who will be recruited in community programs, municipalities, health centers, and social media platforms through phone calls and informational flyers. Those who accept to participate will be informed about the project objectives and procedures. Participation will be voluntary, and everyone will be required to sign the Free and Informed Consent form.

Participants will be allocated into intervention groups: (Boxing training group or Multicomponent training group) or the Control Group (No intervention). The main results will be the physical-functional fitness measured through the Senior Fitness test, Cosmed K5b2, Handgrip strength, ball throw, isokinetic strength, cognitive performance evaluated by neurocognitive and psychological tests, in addition and the risk of falls evaluated by the Biodex® Balance System. Secondary outcomes will be brain activity by means of the electroencephalogram (EEG), bodycomposition, bone mineral density, quality of life and satisfaction with exercise.

The research protocol will follow the CONSORT/SPIRIT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥60 years;
* Community-dwelling older adults;
* Do not present any medical contraindication for physical activity;

Exclusion Criteria:

* Individuals diagnosed with certain disorders or conditions in which exercise is contraindicated such as unstable or ongoing cardiovascular and/or respiratory disorders;
* Presence of major neurological and Neurocognitive disorders (Portuguese version of the Montreal Cognitive Assessment - MoCA) (12);

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Upper Body Power at 3 months and at 6 months, respectively. | Baseline, 6 months
  This will be tested with a 3 kg (Ø 0.60 m) medical ball. Each subject will sit in a chair with the posterior region of the trunk positioned against the back of the chair and hold the ball forward with both hands. Three approved trials will be conducted with one-minute rest intervals between each trial to ensure that fatigue or learning effects do not influence performance. The maximum throwing distance will be determined using a flexible steel tape. Only the best attempt will be used for further analysis (24).
Change from Baseline peak oxygen uptake (VO2 peak) at 6 months | Baseline, 6 months
  Modified Bruce Treadmill Test - This sub-maximal test with incremental protocol including seven stages and performed on a treadmill, standard an open-circuit spirometer technique (Cosmed K5b2, Cosmed, Rome, Italy) will be used.
Change from Baseline Lower-body strength and power at 6 months | Baseline, 6 months
  The knee extensors and flexors will be evaluated using an isokinetic dynamometer (Biodex System 2, USA) at two different angular velocities: 60°/s and 180°/s (22).
Change from Baseline cognitive performance (Inhibition/cognitive flexibility) at 6 months | Baseline, 6 months
  The Stroop Color and Word Test (parameters: words, colors, and words/colors) will be selected to assess response inhibition/cognitive flexibility (14).
Change from Baseline cognitive performance (Processing speed) at 6 months | Baseline, 6 months
  Digit Symbol Substitution Test (DSST, subtest of the Wechsler test of adult intelligence WAIS III) (16, 17) will be used as a measure of high-level information processing speed.
Change from Baseline cognitive performance (Selective recall test) at 6 months | Baseline, 6 months
  Selective recall test [SRT-List A; parameters: consistent long-term recall, long-term storage, delayed recall, and intrusions] to assess verbal learning and multiple-trial memory (14).
Change from Baseline cognitive performance (Verbal short-term memory and verbal working memory) at 6 months | Baseline, 6 months
  The forward digit advancement (DS) test was selected to assess verbal short-term memory and the backward DS to assess verbal working memory (subtest of the Wechsler test of intelligence for adults WAIS III) and total DS score (total DS; calculated by adding forward DS and backward DS) (14, 16).
Change from Baseline cognitive performance (Memory) at 6 months | Baseline, 6 months
  Consortium to establish a registry for the Alzheimer's Disease List Test (CERAD), will be used: word list memory; word list recall; and word list recognition. The parameters: total hits and delayed recall hits (13, 14).
Change from Baseline Psychological testing (Depression) at 6 months | Baseline, 6 months
  The geriatric depression scale (GDS, short version) (18) will be used for depressive symptoms assessment. The GDS-15 evaluates depressive symptoms during the last week and has a dichotomous response scale (Yes/No). On 10 items (2, 3, 4, 6, 8, 9, 10, 12, 14, 15) the answer Yes is rated 1 point and on the remaining items (1, 5, 7, 11, and 13) the answer No is rated 1 point, in the sense that the score indicates presence of depressive symptomatology. The total score of the items is processed by summing the scores on the 15 items, ranging from 0 to 15 points. The 15-item version of the GDS showed the ability to differentiate depressed from nondepressed subjects (18).
Change from Baseline Psychological testing (Anxiety and depression) at 6 months | Baseline, 6 months
  Hospital Anxiety and Depression Scale (HADS) will be used (19). Although the HADS is considered an effective instrument for assessing depressive symptoms in hospital settings, it is a screening measure, and it is of utmost importance to be followed by a psychological assessment. This scale consists of two subscales, one for anxiety and the other for depression. A score between 0 to 7 means absence of depressive or anxious symptoms; a score between 8 to 10 means a possible case of depression or anxiety; and from 11 to 21 as a probable case.
Change from Baseline Psychological testing (Stress) at 6 months | Baseline, 6 months
  Perceived Stress Scale (PSS-10) (20) will be used to assess perceived stress.
Change from baseline on Risk of Falls at 6 months | Baseline, 6 months
  Risk of falls will be evaluated through the Biodex® Balance System (Biodex, Shirley, NY, EUA), using the Fall Risk Test protocol in which the platform is unstable and allows to obtain the risk index and modified version of the Clinical Test of Sensory Interaction and Balance (CTSIB).
Change from baseline on Handgrip strength to 3 and 6 months of exercise and 3-months of follow-up, respectively | Baseline, after 3 months of intervention, 6 months, 3 months follow-up
  The handgrip strength will be measured with a Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA). Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 1 min between them. Three attempts will be made for each hand, using the maximum value of the three registers.
Change from Baseline Brain Activity at 6 months | Baseline, 6 months
  This will be analyzed using an electromyography (EEG) system. All EEG signals will be acquired with the ActiCHamp®, Brain Products,GmbH. With an international 10-20 system with standard 32-channel electrode layout with reference and ground electrodes. The ground will be located on the forehead and the reference will be the Cz channel of the ActiCHamp® equipment. For each participant, the same equipment will be used in all sessions.
Change from baseline Physical-Functional Fitness (upper and lower body strength) at 3 and 6 months of exercise and 3-months of follow-up, respectively | Baseline, after 3 months of intervention, 6 months, 3 months follow-up
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT) (23). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively).
  The chair stand test to assess the strength of the lower body, counting the number of repetitions made in 30s. And the arm curl test to assess the strength on the upper body, using a 3lb (women) and 5lb (men) dumbbell, counting the number of repetitions made in 30s.
Change from baseline Physical-Functional Fitness (8-Foot Up and Go Test) at 3 and 6 months of exercise and 3-months follow-up, respectively. | Baseline, after 3 months of intervention, 6 months, 3 months follow-up.
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT) (23). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively).
  The stand up, walk 8-foot distance (2,44 meters), turn the cone marker around and return to the seated position. The time, in seconds, necessary to complete this test will be registered.
Change from baseline Physical-Functional Fitness (six-minute walk test) at 3 and 6 months of exercise and 3-months follow-up, respectively. | Time Frame: Baseline, after 3 months of intervention, 6 months, 3 months follow-up
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT) (23). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The participants will be asked to walk the longer distance in 6 min time along a corredor.
Change from baseline Physical-Functional Fitness (upper and lower body flexibility) at 3 and 6 months of exercise and 3-months follow-up, respectively. | ime Frame: Baseline, after 3 months of intervention, 6 months, 3 months follow-up
  Physical-functional fitness is going to be measured via the Senior Fitness Test (SFT) (23). This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), agility/dynamic balance (8-foot up-and-go test), aerobic endurance (six-minute walk test) and lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively). The chair sit & reach test to assess the flexibility of the lower body, measured in cm. And the back scratch test to assess flexibility on the upper body, measured in cm.

SECONDARY OUTCOMES:
Sociodemographic Assessments are going to measured at baseline. | Baseline
  Age (years), academic level (primary, secondary, bachelor, master, PhD), civil status (married, separated, widow, single, others), number of medications, diagnosed diseases, falls in the last 12 months.
Change from baseline Quality of Life at 6 months | Baseline, 6 months
  Quality of life will be tested with the World Health Organization Quality of Life Assessment Tool (WHOQOL-Bref).
Change from Baseline Appendicular Skeletal Muscle Mass Index at 6 months | Baseline, 6 months
  Appendicular Skeletal Muscle Mass Index (ASMI), which is the sum of muscle masses of the four limbs described as appendicular skeletal muscle mass adjusted for height (kg/m2), will be analyzed with Dual Energy X-ray Absorptiometry (DXA).
Exercise satisfaction | 6 months
  Will be tested with the physical activity enjoyment scale (PACES) (26). The Portuguese version of the PACES is a validated and reliable instrument to assess enjoyment in group fitness activities. This scale is composed of eight items (e.g., "It is invigorating") preceded by the statement "The physical activity I practice..." to which participants respond through a Likert-type scale with a minimum score of 1 "totally disagree" and maximum score of 7 ("totally agree").
Change from Baseline body mass, fat-free mass, fat mass at 3 and 6 months of exercise and 3-months of follow-up, respectively | Baseline, 3 months, 6 months, 3 months follow-up
  Body mass (kg), fat-free mass (kg) and fat mass (kg) will be analyzed with bioimpedance (InBody 120®).
Change from Baseline Bone Mineral Density at 6 months | Baseline, 6 months.
  They will be analyzed by Dual Energy X-ray Absorptiometry (DXA).

OTHER OUTCOMES:
Change from baseline Caloric Intake at 6 months | Baseline, 6 months
  Caloric intake will be evaluated by a 4-day food record. Macronutrients (i.e., carbohydrate, protein, and fat) will be analyzed as a percentage of total calories consumed.
Exercise intensity | 6 months, during the intervention
  Borg Rating of Perceived Exertion
Applicability of the interventions | 6 months during the intervention
  Adverse events, discomfort or chest pain during training will be measured with the Borg Category ratio scale (CR-10).
Change from baseline Daily Physical Activity levels at 6 months | Baseline, 6 months
  Daily physical activity will be collected with the activity monitors GT3X+ (ActiGraph). Devices are going to be placed on participant´s waist, to measure the activity intensity (counts per minute) during one week. Is addition, physical activity will be also self reported with the IPAQ short version (IPAQ-SV) on the 4 moments of evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Lucimere Bohn, PhD, Principal Investigator — Universidade do Porto; Kessketlen Miranda, PhD student, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Sport, University of Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared. We will only disseminate the results of the study through scientific papers and presentations at scientific conferences

REFERENCES:
- [Background] Santos-Eggimann B, Sirven N. Screening for frailty: older populations and older individuals. Public Health Rev. 2016 Aug 22;37:7. doi: 10.1186/s40985-016-0021-8. eCollection 2016. PMID 29450049
- [Background] Hill NL, Bhargava S, Brown MJ, Kim H, Bhang I, Mullin K, Phillips K, Mogle J. Cognitive complaints in age-related chronic conditions: A systematic review. PLoS One. 2021 Jul 7;16(7):e0253795. doi: 10.1371/journal.pone.0253795. eCollection 2021. PMID 34234373
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Streit IA, Pinto SS, Silva ADS, Bezerra ES. Body weight multicomponent program improves power and functional capacity responses in older adults: A quasi-experimental study. Exp Gerontol. 2021 Nov;155:111553. doi: 10.1016/j.exger.2021.111553. Epub 2021 Sep 14. PMID 34534623
- [Background] Hunter SK, Pereira HM, Keenan KG. The aging neuromuscular system and motor performance. J Appl Physiol (1985). 2016 Oct 1;121(4):982-995. doi: 10.1152/japplphysiol.00475.2016. Epub 2016 Aug 11. PMID 27516536
- [Background] Origua Rios S, Marks J, Estevan I, Barnett LM. Health benefits of hard martial arts in adults: a systematic review. J Sports Sci. 2018 Jul;36(14):1614-1622. doi: 10.1080/02640414.2017.1406297. Epub 2017 Nov 21. PMID 29157151
- [Background] Domingos J, Radder D, Riggare S, Godinho C, Dean J, Graziano M, de Vries NM, Ferreira J, Bloem BR. Implementation of a Community-Based Exercise Program for Parkinson Patients: Using Boxing as an Example. J Parkinsons Dis. 2019;9(3):615-623. doi: 10.3233/JPD-191616. PMID 31282426
- [Background] Shearin S, Braitsch M, Querry R. The effect of a multi-modal boxing exercise program on cognitive locomotor tasks and gait in persons with Parkinson disease. NeuroRehabilitation. 2021;49(4):619-627. doi: 10.3233/NRE-210218. PMID 34806626
- [Background] Combs SA, Diehl MD, Staples WH, Conn L, Davis K, Lewis N, Schaneman K. Boxing training for patients with Parkinson disease: a case series. Phys Ther. 2011 Jan;91(1):132-42. doi: 10.2522/ptj.20100142. Epub 2010 Nov 18. PMID 21088118
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406